CLINICAL TRIAL: NCT02356562
Title: An Open-Label Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of Ombitasvir/ABT-450/Ritonavir (Ombitasvir/ABT-450/r) and Dasabuvir Co-administered With or Without Sofosbuvir (SOF) and Ribavirin (RBV) in Direct-Acting Antiviral Agent (DAA) Treatment-Experienced Adults With Genotype 1 Chronic Hepatitis C Virus (HCV) Infection
Brief Title: A Study of Ombitasvir/Paritaprevir/Ritonavir and Dasabuvir With or Without Sofosbuvir and Ribavirin in Direct-Acting Antiviral Agent Treatment-Experienced Adults With Chronic Hepatitis C Virus Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M14-224
Record Dates: First submitted 2015-02-02; First posted 2015-02-05 (Estimated); Results first posted 2017-11-24 (Actual); Last update posted 2017-12-20 (Actual); Status verified 2017-10

CONDITIONS: Chronic Hepatitis C Infection
Keywords: Hepatitis C; Interferon-Free; Treatment Experienced; Chronic Hepatitis C; Hepatitis C Virus
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic | interventions — ombitasvir; dasabuvir; Viekira Pak; paritaprevir; Sofosbuvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 3-DAA with or without SOF and RBV (Experimental): 3-DAA (ombitasvir/paritaprevir/ritonavir once daily [QD] and dasabuvir twice daily [BID]) with and without sofosbuvir (SOF) QD and with or without ribavirin (RBV) BID for 12 or 24 weeks
  Interventions: Drug: ombitasvir/paritaprevir/ritonavir and dasabuvir; Drug: Sofosbuvir; Drug: Ribavirin

INTERVENTIONS:
Drug: ombitasvir/paritaprevir/ritonavir and dasabuvir — tablet, ombitasvir coformulated with paritaprevir and ritonavir; tablet, dasabuvir
  Other Names: ABT-450/r/ABT-267; Viekira Pak; paritaprevir also known as ABT-450; ombitasvir also known as ABT-267; dasabuvir also known as ABT-333
Drug: Sofosbuvir — tablet
  Other Names: Sovaldi
Drug: Ribavirin — tablet
  Other Names: RBV

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of ombitasvir/paritaprevir/ritonavir and dasabuvir with or without sofosbuvir (SOF) and ribavirin (RBV) in DAA treatment-experienced adults with Genotype 1 Chronic Hepatitis C Virus infection. This study will contain 2 parts.

Part 1: Approximately 20 participants and at least 10 of the 20 participants previously treated with the combination of ombitasvir/paritaprevir/ritonavir and dasabuvir, with or without RBV, and experienced treatment failure.

Part 2: Approximately 10 participants and all participants previously treated with SOF/ledipasvir and experienced treatment failure.

DETAILED DESCRIPTION:
Efficacy, safety, and demographic analyses were performed separately for the 2 study parts using the intent-to-treat (ITT) population, which consists of all enrolled participants who received at least one dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* History of previous direct acting antiviral (DAA) therapy failure; Part 2 only: history of previous direct acting antiviral (DAA) therapy failure and received at least 8 weeks of SOF/ledipasvir; participant must be treatment naïve to all other anti-HCV therapies
* HCV genotype 1 infection
* Females must be post-menopausal, of non-child bearing potential or practicing specific forms of birth control

Exclusion Criteria:

* Positive screen for hepatitis B surface antigen or anti-human immunodeficiency virus antibody
* Discontinuation of the prior DAA treatment for reasons other than virologic failure
* Confirmed presence of hepatocellular carcinoma
* Abnormal lab tests

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-02-03 (Actual); Primary Completion 2016-10-28 (Actual); Study Completion 2017-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Cohen, MD, Study Director — AbbVie

REFERENCES:
- [Derived] King JR, Dutta S, Cohen D, Podsadecki TJ, Ding B, Awni WM, Menon RM. Drug-Drug Interactions between Sofosbuvir and Ombitasvir-Paritaprevir-Ritonavir with or without Dasabuvir. Antimicrob Agents Chemother. 2015 Nov 23;60(2):855-61. doi: 10.1128/AAC.01913-15. Print 2016 Feb. PMID 26596948

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Efficacy, safety, and demographic analyses were performed separately for the 2 study parts using the intent-to-treat (ITT) population, which consists of all enrolled participants who received at least one dose of study drug.
Pre-assignment Details: The intent-to-treat (ITT) population consisted of all enrolled participants who received at least 1 dose of study drug.
Groups:
- Part 1, 3-DAA With SOF With or Without RBV: 3-DAA (ombitasvir/paritaprevir/ritonavir 25 mg/150 mg/100 mg once daily [QD] and dasabuvir 250 mg twice daily [BID]) and sofosbuvir (SOF) 400 mg QD with or without ribavirin (RBV; weight-based dosing 1000 or 1200 mg divided BID or renally adjusted for participants with creatinine clearance < 50 mL/min) for 12 or 24 weeks
- Part 2, 3-DAA With RBV: 3-DAA (ombitasvir/paritaprevir/ritonavir 25 mg/150 mg/100 mg QD and dasabuvir 250 mg BID) with RBV (weight-based dosing 1000 or 1200 mg divided BID or renally adjusted for participants with creatinine clearance < 50 mL/min) for 24 weeks
Period: Overall Study
Arm/Group | Part 1, 3-DAA With SOF With or Without RBV | Part 2, 3-DAA With RBV
Started | 22 | 7
Completed | 20 | 6
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Re-entered treatment in a previous study | 1 | 0
Not completed — site closure | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1, 3-DAA With SOF With or Without RBV | Part 2, 3-DAA With RBV | Total
Number analyzed (Participants) | 22 | 7 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (6.41) | 65.3 (9.60) | NA (NA) — Per protocol, data from Parts 1 and 2 were not combined for analysis.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 1 | 8
  Male | 15 | 6 | 21

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Part 1 Participants With Sustained Virologic Response 12 (SVR12) Weeks Posttreatment
Description: SVR12 was defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) level less than the lower limit of quantification [<LLOQ]) 12 weeks after the last dose of study drug.
Time Frame: 12 weeks after the last dose of active drug
Population: All Part 1 participants who received at least 1 dose of study drug (ITT population). Per protocol, data from Parts 1 and 2 were not combined for analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1, 3-DAA With SOF With or Without RBV
Number analyzed (Participants) | 22
percentage of participants | 95.5 [78.2 to 99.2]

2. Secondary Outcome: Percentage of Part 2 Participants With Sustained Virologic Response 12 (SVR12) Weeks Post-treatment
Description: SVR12 was defined as plasma HCV RNA level <LLOQ 12 weeks after the last dose of study drug
Time Frame: 12 weeks after the last dose of active drug
Population: All Part 2 participants who received at least 1 dose of study drug (ITT population). Per protocol, data from Parts 1 and 2 were not combined for analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2, 3-DAA With RBV
Number analyzed (Participants) | 7
percentage of participants | 85.7 [48.7 to 97.4]

3. Secondary Outcome: Percentage of Participants With On-treatment Virologic Failure
Description: On-treatment virologic failure was defined as confirmed HCV RNA ≥ LLOQ after < LLOQ during treatment, confirmed increase of > 1 log (subscript)10(subscript) IU/mL above the lowest post-baseline HCV RNA during treatment, or HCV RNA ≥ LLOQ persistently during treatment with at least 6 weeks of treatment.
Time Frame: Up to week 24
Population: All participants who received at least 1 dose of study drug (ITT population). Per protocol, data from Parts 1 and 2 were not combined for analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1, 3-DAA With SOF With or Without RBV | Part 2, 3-DAA With RBV
Number analyzed (Participants) | 22 | 7
percentage of participants | 0.0 [0.0 to 14.9] | 14.3 [2.6 to 51.3]

4. Secondary Outcome: Percentage of Participants With Post-Treatment Relapse
Description: Post-treatment relapse was defined as confirmed HCV RNA ≥ LLOQ between end of treatment and 12 weeks after the last dose of study drug among participants completing treatment and with HCV RNA < LLOQ at the end of treatment.
Time Frame: Within 12 weeks after the last actual dose of active study drug
Population: All participants who received at least 1 dose of study drug (ITT population) with HCV RNA < LLOQ at the end of treatment and completed treatment. Per protocol, data from Parts 1 and 2 were not combined for analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1, 3-DAA With SOF With or Without RBV | Part 2, 3-DAA With RBV
Number analyzed (Participants) | 21 | 6
percentage of participants | 4.8 [0.8 to 22.7] | 0.0 [0.0 to 39.0]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from the time of study drug administration until 30 days after the last dose of study drug (up to 28 weeks).
Description: TEAEs and TESAEs are defined as any adverse event (AE) with an onset date that is on or after the date of the first dose of study drug until 30 days after the last dose of study drug and were collected whether elicited or spontaneously reported by the participant.
Groups:
- Part 1, 3-DAA With SOF With or Without RBV: 3-DAA (ombitasvir/paritaprevir/ritonavir [25 mg/150 mg/100 mg once daily [QD] and dasabuvir [250 mg twice daily [BID]) and sofosbuvir (SOF) 400 mg QD with or without ribavirin (RBV; weight-based dosing 1000 or 1200 mg divided BID or renally adjusted for participants with creatinine clearance < 50 mL/min) for 12 or 24 weeks.
- Part 2, 3-DAA With RBV: 3-DAA (ombitasvir/paritaprevir/ritonavir [25 mg/150 mg/100 mg QD and dasabuvir [250 mg BID) with RBV (weight-based dosing 1000 or 1200 mg divided BID or renally adjusted for participants with creatinine clearance < 50 mL/min) for 24 weeks.
Arm/Group | Part 1, 3-DAA With SOF With or Without RBV | Part 2, 3-DAA With RBV
Serious Adverse Events (participants affected / at risk) | 2/22 | 0/7
Other Adverse Events (participants affected / at risk) | 20/22 | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1, 3-DAA With SOF With or Without RBV (N=22) | Part 2, 3-DAA With RBV (N=7)
CELLULITIS (Infections and infestations) | 1 | 0
PNEUMONIA (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1, 3-DAA With SOF With or Without RBV (N=22) | Part 2, 3-DAA With RBV (N=7)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 1
HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 1 | 0
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 1 | 0
VERTIGO (Ear and labyrinth disorders) | 1 | 0
VERTIGO POSITIONAL (Ear and labyrinth disorders) | 1 | 0
CUSHING'S SYNDROME (Endocrine disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 0
DENTAL CARIES (Gastrointestinal disorders) | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 4 | 1
DRY MOUTH (Gastrointestinal disorders) | 1 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 | 1
IMPAIRED GASTRIC EMPTYING (Gastrointestinal disorders) | 0 | 1
MOUTH ULCERATION (Gastrointestinal disorders) | 1 | 0
NAUSEA (Gastrointestinal disorders) | 3 | 0
ORAL PAIN (Gastrointestinal disorders) | 1 | 0
VOMITING (Gastrointestinal disorders) | 1 | 0
ASTHENIA (General disorders) | 2 | 0
CYST (General disorders) | 1 | 0
ENERGY INCREASED (General disorders) | 1 | 0
FATIGUE (General disorders) | 7 | 3
FEELING COLD (General disorders) | 1 | 0
MALAISE (General disorders) | 0 | 1
OEDEMA PERIPHERAL (General disorders) | 1 | 0
PYREXIA (General disorders) | 2 | 0
CONJUNCTIVITIS BACTERIAL (Infections and infestations) | 0 | 1
EAR INFECTION (Infections and infestations) | 1 | 0
GASTROENTERITIS (Infections and infestations) | 2 | 0
INFLUENZA (Infections and infestations) | 1 | 0
SINUSITIS (Infections and infestations) | 1 | 0
STAPHYLOCOCCAL SKIN INFECTION (Infections and infestations) | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 2 | 0
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 1 | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 1
CREATININE RENAL CLEARANCE DECREASED (Investigations) | 1 | 1
GLUCOSE TOLERANCE IMPAIRED (Metabolism and nutrition disorders) | 0 | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 | 0
INCREASED APPETITE (Metabolism and nutrition disorders) | 1 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
OSTEOPENIA (Musculoskeletal and connective tissue disorders) | 1 | 0
DIZZINESS (Nervous system disorders) | 3 | 0
HEADACHE (Nervous system disorders) | 8 | 1
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 | 0
SYNCOPE (Nervous system disorders) | 1 | 0
AGITATION (Psychiatric disorders) | 1 | 0
EUPHORIC MOOD (Psychiatric disorders) | 1 | 0
INSOMNIA (Psychiatric disorders) | 4 | 0
IRRITABILITY (Psychiatric disorders) | 2 | 0
HYPERTONIC BLADDER (Renal and urinary disorders) | 1 | 0
MENOPAUSAL SYMPTOMS (Reproductive system and breast disorders) | 1 | 0
PROSTATITIS (Reproductive system and breast disorders) | 1 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 | 0
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 2 | 0
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ECZEMA (Skin and subcutaneous tissue disorders) | 0 | 1
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 | 0
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 1 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 1 | 0
RASH (Skin and subcutaneous tissue disorders) | 2 | 0
SKIN LESION (Skin and subcutaneous tissue disorders) | 0 | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 | 0
FLUSHING (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.